CLINICAL TRIAL: NCT05927181
Title: Flapless Immediate Implants in Type 1 Alveoli: Soft Tissue Alterations Following a Trimodal Approach With or Without Modifying Osseous and Mucosal Compartments (TAOM vs TA) in the Aesthetic Zone: A Comparative Prospective Study.
Brief Title: Immediate Implants: to Graft or Not to Graft, That is the Question.
Acronym: TAOM-TA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMA-USE-001
Record Dates: First submitted 2023-05-19; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Dental Implant
Keywords: Immediate Implants; soft tissue graft; immediate implant restoration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodal Approach with Osseous and Mucosal compartment modification: TAOM (Experimental): Flapless immediate implant placement and provisional restoration with alveolar filling and connective tissue graft.
  Interventions: Procedure: TAOM
- Trimodal Approach: TA (Active Comparator): Flapless immediate implant placement and provisional restoration.
  Interventions: Procedure: TAOM

INTERVENTIONS:
Procedure: TAOM — In the TAOM group, the gap between the implant and the facial bone wall was grafted with inorganic bovine bone (Geistlich Bio-Oss®; Geistlich Pharma AG, Wolhusen, Switzerland) and, in addition, a connective tissue graft (CTG) was placed submucosally on the labial bone plate by means of an envelope technique.
  Other Names: Trimodal approach with osseous and mucosal interventions.

SUMMARY:
The aim was to compare two protocols for immediate implants with fixed provisional restoration, no grafting (trimodal approach=TA) versus grafting both osseous gap and peri-implant mucosa (trimodal approach with modification of the osseous and mucosal compartments =TAOM) by measuring the soft tissue changes overtime. The periodontal phenotype was registered, to investigate a relationship between its thickness and the clinical outcomes.

DETAILED DESCRIPTION:
The study protocol was approved by the CEIm Quiron Salud Catalunya institutional research ethic committee (Approval code:2022/102_MAX:CEX). This prospective clinical study includes patients who were enrolled and treated in two private practices (GC and JGF). All eligible patients were consecutively selected for two study groups receiving immediately placed flapless implants and the provisional restoration. Patients were informed about the characteristics of the study and signed their informed consent before the study began.

Patient population

Patients in need of single implant supported restorations in the anterior maxilla (canines, lateral and central incisors) were selected for this study. The indications for tooth extractions were cavities, endodontic complications (e.g., root fracture), internal resorption and prosthetic reasons. The patients had to fulfil the following inclusion and exclusion criteria:

Inclusion criteria:

* ≥18 years of age
* Need for tooth extraction in the anterior maxilla (13-23) due to cavities, internal resorption, fractures, restorative problems, endodontic complications and prosthetic reasons.
* The failing tooth has adjacent and opposing natural teeth
* Adequate oral hygiene (Bleeding on probing <20%; Plaque index <20%);
* Absence of active and uncontrolled periodontal disease
* Sufficient mesial-distal and interocclusal space for implant placement and definitive restoration
* Sufficient interocclusal space to design a non-occluding provisional restoration

Exclusion criteria:

* Systemic metabolic or osseous disease that could compromise peri-implant tissue healing
* Acute infection in the treatment area
* Absence of one or both adjacent teeth
* Non-integrity of the buccal bone wall (dehiscence or fenestration) observed during surgery, or when tooth extraction has altered the integrity of the osseous and gingival architecture

The participants were screened by two investigators (GC & JGF) and comprised two consecutive study groups with the following interventions:

1. Flapless immediate implant placement and provisional restoration (trimodal approach: TA) (n=15).
2. Flapless immediate implant placement and provisional restoration with alveolar filling and connective tissue graft (trimodal approach with osseous and mucosal compartment modification: TAOM) (n=16).

Treatment protocol and follow-up

Four visits were intended to be delivered in each participant. Following the selection of candidates, study casts were prepared for all patients as well as preoperative photographs and parallel periapical radiographs of the problematic tooth. Rigid stents were prepared with light-cured resin, covering the incisal edges of at least one adjacent tooth on each side of the target tooth. Measurements from reference points to mid-buccal soft tissue height and mesial and distal papillae were recorded at T0. The stents were > 2 mm thick so they could be modified to allow for a perfect fit over the final restoration.

All surgical procedures were performed by two experienced surgeons and investigators (GC& JGF). Without raising a mucoperiosteal flap, a careful tooth extraction was performed, allowing for the preservation of soft and hard tissues. In 10 patients, the Benex Extractor® (Benex Root Extraction System, Hager and Meisinger GMbH, Neuss, Germany) was used to ensure atraumatic extraction. Then, a detailed examination of the buccal bone wall was carried out to verify its integrity. In the cases when the integrity of the bone wall was in question, the patient was excluded from the study and the implant was placed by means of conventional protocols.

Measurement of the total periodontal thickness (phenotype) was taken at this time by means of an analogic calliper located 5 mm apical to the buccal gingival margin, to locate the bundle bone level.

Then, the implant bed was prepared on the palatal side of the extraction socket in accordance with the manufacturer's instructions (Bone Level -BL- and Tissue Level -TL-, Straumann AG, Switzerland; Thoma et al., 2021). The implant was placed securing the ideal position at a depth of 2mm for the TL implant and 4mm for the BL implant and in a palatal position allowing for a direct screw-retained restoration (1-3 mm from the bone wall) for all implants. It was also verified that the wall of the post-extraction socket was not perforated during implant bed preparation. The implant had to show good primary stability in its ideal position, in order to avoid being excluded from the study. In the TA group, no material was used to fill the gap between the implant and the osseous wall and no soft tissue graft was attempted either. In the TAOM group, the gap between the implant and the facial bone wall was grafted with inorganic bovine bone (Geistlich Bio-Oss®; Geistlich Pharma AG, Wolhusen, Switzerland) and, in addition, a connective tissue graft (CTG) was harvested from the anterior palate region and placed submucosally on the labial bone plate by means of an envelope technique.

Following implant placement, an acrylic resin implant-supported provisional restoration was prepared, adapted and delivered for all implants. All provisional restorations were directly screw-retained and designed with no occlusal contacts, neither in maximum intercuspal position nor in excursive movements. The emergence profile was mainly flat or concave in interproximal and palatal sides, and slightly convex in the buccal aspect to support the soft tissues for the TA group. In the TAOM group, it was slightly concave to provide space for the soft-tissue graft and avoid isquemia in the marginal mucosa. Intra-oral radiographs were taken to check implant position and the fit of the restoration. Systemic antibiotics (Azitromicin-500mg/24h/3days) and anti-inflammatories (Dexketoprofen-25mg/8h/3days) were prescribed, together with a clorhexidine 0.20 % gel twice a day for one week. Patients were then recalled for a post-operative check-up and sutures were removed after 14 days.

At 3 months, final impressions were made. After abutment selection and bisque try-ins, final restorations were permanently placed at 4 months.

The tooth-supported acrylic resin measuring stent was then adapted to allow for a complete fit on the incisal edges of both neighbouring teeth, to ensure a reliable positioning and measurement reference.

The first measurement was at day 0 (Immediate implant placement and provisionalisation). Patient recall appointments for examinations and measurements took place at 3, 6 and 12 months. No activities were performed to increase compliance or adherence in the selected patients beyong compliance of a good clinical practice.

Outcome measures The primary outcome variable of this study was the vertical midfacial soft tissue change from baseline (before tooth extraction) to 12 months following implant placement.

The secondary outcome measures were mesial and distal papillae vertical changes, periodontal phenotype at implant site, and mechanical complications.

The clinical outcomes were measured as follows:

* Vertical soft tissue changes were calculated through the distance from reference measuring points on the stent to mesial (MP) and distal (DP) papillae, and gingival zenith (Z) of the implant restoration. Distances were measured by means of a precision digital calliper that can display measurements as small as tenths of a millimetre. Three dimples were marked in the stent, in approximately the vertical projection of papillae and zenith (Supplementary figure 1a). Measurements were taken before tooth extraction (baseline) T0 and at 3 (T3), 6 (T6) and 12 (T12) months following the intervention.
* Periodontal phenotype thickness was measured by means of an analogical calliper that was able to show tenths of a millimetre. It was located 5 mm apical to the buccal gingival margin immediately after tooth extraction.
* Mechanical complications were assessed and included: screw loosening, loss of retention, chipping of acrylic or porcelain complications.

ELIGIBILITY:
Inclusion Criteria:

* Need for tooth extraction in the anterior maxilla (13-23) due to cavities, internal resorption, fractures, restorative problems, endodontic complications and prosthetic reasons.
* The failing tooth has adjacent and opposing natural teeth
* Adequate oral hygiene (Bleeding on probing <20%; Plaque index <20%);
* Absence of active and uncontrolled periodontal disease
* Sufficient mesial-distal and interocclusal space for implant placement and definitive restoration
* Sufficient interocclusal space to design a non-occluding provisional restoration

Exclusion Criteria:

* Systemic metabolic or osseous disease that could compromise peri-implant tissue healing.
* Acute infection in the treatment area
* Absence of one or both adjacent teeth
* Non-integrity of the buccal bone wall (dehiscence or fenestration) observed during surgery, or when tooth extraction has altered the integrity of the osseous and gingival architecture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Distance from measuring points on the reference stent to gingival zenith of the implant restoration in tenths of a milimetre by means of a precision digital calliper. | 12 months
  Vertical midfacial soft tissue change from baseline (before tooth extraction) to 12 months following implant placement.

SECONDARY OUTCOMES:
Distance from measuring points on the reference stent to mesial and distal papillae of the implant restoration in tenths of a milimetres by means of a precision digital calliper. | 12 months
  Vertical mesial and distal papillae soft tissue change from baseline (before tooth extraction) to 12 months following implant placement.
Periodontal thickness at 5mm apical to the gingival margin in tenths of a milimetre. | Baseline
  Thickness at implant site at 5 mm apical to the buccal gingival margin from the external queratinized tissue to internal part of the buccal bundle bone.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo G Cabello, Principal Investigator — Private Practice, Málaga, Spain; Javier J Fabrega, Principal Investigator — Private Practice, Madrid, Spain
Locations (1):
- Maria Del Rosario Rioboo Crespo, Madrid, Spain